CLINICAL TRIAL: NCT04877600
Title: The Relationship Between Cognitive and Motor Functions, and Dual Task Performance in Community Dwelling Older Adults: Gender Differences
Brief Title: Dual Task Performance in Community Dwelling Older Adults
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, AYŞE ÜNAL, PT.,PhD, Pamukkale University
Other Study IDs: 60116787-020/77265
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Dual Task; Community Dwelling Older Adult
Keywords: dual task; community dwelling older adult; motor performance; cognitive status

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- gender difference: dual task performance
  Interventions: Other: dual task performance

INTERVENTIONS:
Other: dual task performance — dual task performance measurement

SUMMARY:
Dual task performances may be impaired with the impairment in motor performance and cognitive functions due to aging. The aim of the present study is to investigate the gender differences in dual task performance. A total of 82 community dwelling older adults (41 males and 41 females) aged between 65 and 75 years were included in the study. Motor performance was evaluated with sit-to-stand test, the timed up and go test, 10 m walking test and cognitive functions were evaluated with Montreal Cognitive Assessment Test. Dual task performances were evaluated as motor-motor and cognitive-motor performance.

ELIGIBILITY:
Inclusion Criteria:

* The individuals aged between 65 and 75 years, who agreed for participation, who received 8 or higher points from Hodkinson Mental test, who had no neurologic/orthopedic problems that could affect balance and walking, or communication problem were included in the study.

Exclusion Criteria:

* The individuals who were using 3 or more medications that could affect motor and cognitive functions, and the ones who could not complete the tests were excluded.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — A total of 82 healthy community dwelling older adults (41 males and 41 females) aged between 65 and 75 years
Study Population: Dual task performances may be impaired with the impairment in motor performance and cognitive functions due to aging. Because of this, we aimed to investigate the gender differences in dual task performance.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Dual Task Performance | 5 minutes
  Assessment of Dual Task Performance

SECONDARY OUTCOMES:
Montreal Cognitive Assessment Scale | 5 minutes
  Assessment of Cognitive Functions
Timed Up and Go | 5 minutes
  Assessment of Physical Performance
30 Seconds Sit-to-Stand Test | 5 minutes
  Assessment of Physical Performance
10 Meter Walking Test | 5 minutes
  Assessment of Physical Performance

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No